CLINICAL TRIAL: NCT00156377
Title: Investigation of the Influence of Intranasal Mupirocin on the Prevalence of S. Aureus Nosocomial Infections by Eradication of Intranasal S. Aureus
Brief Title: Prophylaxis With Intranasal Mupirocin for Prevention of S. Aureus Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4710F-186
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2005-09

CONDITIONS: Cross Infection; Staphylococcal Infections
Keywords: Mupirocin; Staphylococcus aureus; Nasal Cavity; Preventive measures
MeSH Terms: conditions — Cross Infection; Staphylococcal Infections | interventions — Mupirocin

INTERVENTIONS:
Drug: Mupirocin

SUMMARY:
In order to evaluate the effect of eliminating nasal carriage by mupirocin prophylaxis on subsequent Staphylococcus aureus infection, a prospective randomized trial was performed particularly including patients with predisposing risk factors for S. aureus infections.

DETAILED DESCRIPTION:
In a past study, we showed that there is a strong correlation between strains colonizing the anterior nares, strains isolated from the presumed foci of infection, and strains isolated from blood in patients with Staphylococcus aureus bacteremia. These results suggested that a substantial proportion of cases of systemic S. aureus infections appear to be of endogenous origin and that eradication of nasal colonization should be the chief strategy for reducing the incidence of hospital-acquired S. aureus infections.

In order to evaluate the effect of eliminating nasal carriage by mupirocin prophylaxis on subsequent S. aureus infection, a prospective randomized trial was performed particularly including patients with predisposing risk factors for S. aureus infections. All patients admitted to selected units in clinics for anaesthesiology, hemato-oncology, cardiac surgery, and orthopedics at the University Hospital of Muenster were regularly screened for nasal carriage, i.e. at admission and, subsequently, on a weekly basis. S. aureus carrying patients were prospectively randomized, to be either treated with mupirocin for 5 days, or left untreated. Patients infected with S. aureus at admission and patients detected to be MRSA carrier were excluded from randomization.

Patients were regularly seen during the course of their hospital stay and predisposing/conditional risk factors were systematically documented. In both groups (untreated patients and patients with mupirocin prophylaxis), all nosocomial infections were documented according to CDC guidelines. If infected, specimens were taken for microbiological diagnosis. All S. aureus isolates (from the anterior nares as well as from the focus of infection) were collected and were genotyped.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to selected units in clinics for anaesthesiology, hemato-oncology, cardiac surgery, and orthopedics at the University Hospital of Muenster (following information on the study and agreement of the patient).

Exclusion Criteria:

* Patients infected with S. aureus at admission
* S. aureus infection within 48 hours following admission
* Patients detected to be carrier of Methicillin-resistant S. aureus
* Hospital stay shorter than 72 hours
* Patients with anatomic abnormalities in the anterior nares
* Allergy or hypersensitivity to mupirocin or other substances of the nasal ointment
* Persons younger than 18 years
* Known pregnancy
* Persons with psychiatric diseases
* Persons with limited contractual capability and judiciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2002-11

PRIMARY OUTCOMES:
Staphylococcus aureus infection any time after 5 days of mupirocin ointment

SECONDARY OUTCOMES:
Presence or abscence of risk factors associated with S. aureus infections at any time during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Christof von Eiff, MD, Principal Investigator — University Hospital of Muenster, Institute of Medical Microbiology
Locations (1):
- Institute of Medical Microbiology, University Hospital of Muenster, Münster, Germany

REFERENCES:
- [Background] von Eiff C, Becker K, Machka K, Stammer H, Peters G. Nasal carriage as a source of Staphylococcus aureus bacteremia. Study Group. N Engl J Med. 2001 Jan 4;344(1):11-6. doi: 10.1056/NEJM200101043440102. PMID 11136954
- [Background] von Eiff C, Kipp F, Becker K. Intranasal mupirocin to prevent postoperative infections. N Engl J Med. 2002 Oct 10;347(15):1207-8; author reply 1207-8. doi: 10.1056/NEJM200210103471518. No abstract available. PMID 12374887
- See also: Home page of the Institute of Medical Microbiology of the University Hospital of Muenster — http://mibi1.uni-muenster.de/